CLINICAL TRIAL: NCT00665223
Title: A Multicentre, Multinational, Randomised, Double-Blind, Parallel-Group Study Comparing ACR16 45 mg Once-Daily or Twice-Daily Versus Placebo for the Symptomatic Treatment of Huntington's Disease
Brief Title: A Study of Treatment With Pridopidine (ACR16) in Participants With Huntington's Disease
Acronym: MermaiHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACR16 C008
Record Dates: First submitted 2008-04-22; First posted 2008-04-23 (Estimated); Results first posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-07

CONDITIONS: Huntington's Disease
Keywords: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — pridopidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive a placebo capsule matching to ACR16 once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 26), placebo capsule will be taken twice daily as 2 separate doses.
  Interventions: Drug: Placebo
- ACR16 45 mg (Experimental): Participants will receive ACR16 45 milligrams (mg) capsule orally once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 26), one ACR16 45 mg capsule and one placebo capsule will be taken as 2 separate doses.
  Interventions: Drug: ACR16; Drug: Placebo
- ACR16 90 mg (Experimental): Participants will receive ACR16 45 mg capsule once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 26), ACR16 45 mg capsule will be taken twice daily as 2 separate doses (total dose: 90 mg)
  Interventions: Drug: ACR16

INTERVENTIONS:
Drug: ACR16 — Capsules will be swallowed whole with water.
  Other Names: Pridopidine
  Arms: ACR16 45 mg; ACR16 90 mg
Drug: Placebo — Capsules will be swallowed whole with water.
  Arms: ACR16 45 mg; Placebo

SUMMARY:
The purpose of this study is to determine if ACR16 is effective and safe in the symptomatic treatment of Huntington's disease.

DETAILED DESCRIPTION:
The primary objective in the present study is to confirm whether ACR16 is efficacious in improving voluntary motor function in Huntington's disease based on the Unified Huntington"s Disease Rating Scale (UHDRS) subscale. These symptoms seem to be most important for the functional disability associated with the disorder. To achieve this, participants are randomized to ACR16 45 mg once daily, ACR16 45 mg twice daily, or placebo treatment in equal proportions in a parallel design for a treatment duration of 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written Informed Consent prior to any study related procedure.
* Huntington's disease diagnosed with the aid of clinical features and a positive family history and/or the presence of ≥ 36 CAG repeats in the Huntington gene.
* Male or female age ≥ 30 years.
* Willing and able to take oral medication and able to comply with the study specific procedures.
* Ambulatory, being able to travel to the assessment centre, and judged by the Investigator as likely to be able to continue to travel for the duration of the study.
* Availability of a caregiver or family member to accompany the participant.
* A sum of ≥ 10 points on the mMS at the screening visit.
* For participants taking allowed antipsychotic medication, the dosing of medication must have been kept constant for at least 6 weeks before randomization. The allowed antipsychotic medication is Amisulpride, Haloperidol, Olanzapine, Risperidone, Sulpiride, or Tiapride.
* For participants taking allowed antidepressant or other psychotropic medication, the dosing of medication must have been kept constant for at least 6 weeks before randomization.
* Willing to provide a blood sample for CAG analysis (where CAG result is not already available).
* In France only, the participant must be affiliated to a social security system or be a beneficiary of such a system.

Exclusion Criteria:

* Unable to give written informed consent.
* Treatment with any non-allowed antipsychotic medication within 12 weeks of randomization. The non-allowed antipsychotic medication is any medication other than Amisulpride, Haloperidol, Olanzapine, Risperidone, Sulpiride, or Tiapride.
* Treatment with the antidepressants Fluoxetine or Paroxetine within 6 weeks of randomization.
* Use of Tetrabenazine within 12 weeks of randomization, or at any time during the study period.
* Treatment with any investigational product within 4 weeks of randomization.
* Use of tricyclic antidepressants, class I antiarrhythmics, and strong CYP2D6 inhibitors such as Ajmalicine, Chinidin/Quinidine and Ritonavir, within 6 weeks of randomization.
* Participants previously included into this study.
* A prolonged QTc interval at screen (defined as a QTc interval of > 450 milliseconds [msec] for males or > 470 msec for females), or other clinically significant heart conditions.
* Creatinine clearance <40 milliliters (mL)/minute (min) as measured at the screening visit.
* Any clinically significant, abnormal, baseline laboratory result which in the opinion of the Investigator, affects the participants' suitability for the study or puts the participant at risk if he/she enters the study.
* Clinically significant hepatic or renal impairment.
* Participants with a history of epilepsy or a history of seizure(s) of unknown cause.
* Severe intercurrent illness, which, in the opinion of the Investigator, may put the participant at risk when participating in the trial or may influence the results of the trial or affect the participants' ability to take part in the trial.
* Alcohol and/or drug abuse as defined by Diagnostic and Statistical Manual - Fourth Edition - Text Revision (DSM IV-TR) criteria for substance abuse - this includes the illicit use of cannabis within the last 12 months.
* Participants with suicidal ideation, defined as a positive score on criteria for major depressive episode, item A9 on the DSM-IV-TR criteria for a Major Depressive Episode.
* Females who are pregnant or lactating.
* Females who are of child bearing potential and not taking adequate contraceptive precautions are excluded from the trial. Females of child bearing potential taking acceptable contraceptive precautions can be included.
* Known allergy to any ingredients of the trial medication or placebo.
* Any previous participation in a clinical study with ACR16.
* Participants currently receiving deep brain stimulation.
* Participants with a history of surgical procedures aiming to improve the symptoms of Huntington's disease, such as neural transplantations, lesions of the central nervous system, infusions of neurotrophic agents or previous attempts of deep brain stimulation.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2008-04-24 (Actual); Primary Completion 2010-06-14 (Actual); Study Completion 2010-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (31):
- Austria (2):
  - LKH -Univ. Klinikum Graz, Universitaetsklinik fur Psychiatrie Graz, Graz, Styria
  - Innsbruck Medical University, Anichstraße 35, Innsbruck, Tyrol
- University Hospital Gasthuisberg, Leuven, Flemish Brabant, Belgium
- France (4):
  - CHU Roger Salengro, Lille, Hauts-de-France
  - Hôpital Purpan, Place Docteur-Baylac, Bâtiment F, Toulouse, Midi-Pyrénées Region
  - Hôpital Nord, CHU d'Amiens, Service de Neurologie, Amiens, Picardie
  - CHU La Timone, 264 Rue Saint Pierre, Marseille, Provence-Alpes-Côte d'Azur Region
- Germany (7):
  - Universitätsklinik Ulm, Neurologie/ Oberer Eselberg 45/1, Ulm, Baden-Wurttemberg
  - Klinikum rechts der Isar der Technischen Universität München, Neurologische Klinik und Poliklinik, Ismaninger Str. 22, München, Bavaria
  - Isar Amper Klinikum gemeinnützige GmbH, Klinik Taufkirchen (Vils), Bräuhausstr.5, Taufkirchen (Vils), Bavaria
  - St. Josef Hospital, Ruhr University Bochum, Gudrunstraße 56, Bochum, North Rhine-Westphalia
  - Westfaelische Wilhelms-Universitaet Muenster, Klinik fur Neurologie, Münster, North Rhine-Westphalia
  - Universitat Dresden, Klinikum Carl Gustav Carus, Fetscherstr. 74, Dresden, Saxony
  - Klinik für Psychiatrie und Psychotherapie, Charité - Universitätsmedizin Berlin, Schumannstrasse 20/21, Berlin
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale Neurologico "Carlos Besta", Department of Movement Disorders, 11 via Celoria, Milan, Lombardy
  - IRCCS Neuromed, Localita Camarelle, Pozzilli, Molise
- Portugal (2):
  - University Hospital of Coimbra, Av. Rissaya Barreto, Coimbra, Baixo Mondego
  - Centro de Estudos Egas Moniz, Faculdade de Medicina de Lisboa, Av. Prof. Egas Moniz, Lisbon
- Spain (4):
  - Hospital Mútua de Terrassa, C/ Castell, Terrassa, Catalonia
  - Hospital Clinic of Barcelona, Calle Villarroel, 170, Barcelona
  - Hospital Ramon y Cajal, Carretera Colemenar km 9.100, Madrid
  - Hospital Universitario La Fe, Avda. Campanar 21,, Valencia
- United Kingdom (9):
  - R&D Headquarters, Barberry Centre, 25 Vincent Drive, Birmingham, England/West Midlands
  - Department of Clinical Genetics, St Mary's Hospital, Hathersage Road, Manchester, North West England
  - First Floor Argyll House, Fosterhill, Cornhill Road, Aberdeen, Scotland
  - SE Scotland Genetic Service, Western General Hospital, Crewe Road, Edinburgh, Scotland
  - Churchill Hospital, Old Road, Headington, Oxford, South East England
  - Academic Neurology Unit, E Floor Medical School Beech Hill Road, Sheffield, South Yorkshire
  - Institute of Human Genetics, Centre for Life, Central Parkway, Newcastle upon Tyne, Tyne and Wear
  - Cardiff University School of Medicine, Department of Neurology & Medical Genetics, Heath Park, Cardiff, Wales
  - Cambridge Centre for Brain repair, Cambridge University, Cambridge

REFERENCES:
- [Derived] Darpo B, Geva M, Ferber G, Goldberg YP, Cruz-Herranz A, Mehra M, Kovacs R, Hayden MR. Pridopidine Does Not Significantly Prolong the QTc Interval at the Clinically Relevant Therapeutic Dose. Neurol Ther. 2023 Apr;12(2):597-617. doi: 10.1007/s40120-023-00449-w. Epub 2023 Feb 22. PMID 36811812
- [Derived] de Yebenes JG, Landwehrmeyer B, Squitieri F, Reilmann R, Rosser A, Barker RA, Saft C, Magnet MK, Sword A, Rembratt A, Tedroff J; MermaiHD study investigators. Pridopidine for the treatment of motor function in patients with Huntington's disease (MermaiHD): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2011 Dec;10(12):1049-57. doi: 10.1016/S1474-4422(11)70233-2. Epub 2011 Nov 7. PMID 22071279

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants that completed the randomized phase to week 26 on-treatment were given the option to continue treatment in the open-label phase.
Groups:
- Placebo/ACR16 90 mg: Randomized phase: Participants received a placebo capsule matched to ACR16 once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 26), placebo capsule was taken twice daily as 2 separate doses.
  Open-label phase: Participants received ACR16 45 milligrams (mg) capsule once daily for the first 4 weeks (Weeks 26 to 30). After 4 weeks (Weeks 31 to 52), ACR16 45 mg capsule was taken twice daily as 2 separate doses (total dose: 90 mg).
- ACR16 45 mg/90 mg: Randomized phase: Participants received ACR16 45 mg capsule orally once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 26), one ACR16 45 mg capsule and one placebo capsule were taken as 2 separate doses.
  Open-label phase: Participants received ACR16 45 mg capsule once daily for the first 4 weeks (Weeks 26 to 30). After 4 weeks (Weeks 31 to 52), ACR16 45 mg capsule was taken twice daily as 2 separate doses (total dose: 90 mg).
- ACR16 90 mg/90 mg: Randomized Phase: Participants received ACR16 45 mg capsule once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 26), ACR16 45 mg capsule was taken twice daily as 2 separate doses (total dose: 90 mg).
  Open-label phase: Participants received ACR16 45 mg capsule once daily for the first 4 weeks (Weeks 26 to 30). After 4 weeks (Weeks 31 to 52), ACR16 45 mg capsule was taken twice daily as 2 separate doses (total dose: 90 mg).
Period: Randomized Phase (26 Weeks)
Arm/Group | Placebo/ACR16 90 mg | ACR16 45 mg/90 mg | ACR16 90 mg/90 mg
Started | 144 | 148 | 145
Received at Least 1 Dose of Study Drug | 144 | 148 | 145
Completed | 126 | 136 | 124
Not Completed | 18 | 12 | 21
Not completed — Adverse Event | 13 | 9 | 15
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 2 | 3
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Other than specified | 0 | 0 | 1
Period: Open-Label Period (26 Weeks)
Arm/Group | Placebo/ACR16 90 mg | ACR16 45 mg/90 mg | ACR16 90 mg/90 mg
Started | 113 | 125 | 115
Completed | 97 | 108 | 100
Not Completed | 16 | 17 | 15
Not completed — Adverse Event | 8 | 11 | 7
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 1 | 2
Not completed — Withdrawal by Subject | 5 | 3 | 4
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Other than specified | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug and had undergone at least 1 clinical assessment post randomization.
Groups:
- Placebo/ACR16 90 mg: Randomized-phase: Participants received a placebo capsule matched to ACR16 once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 26), placebo capsule was taken twice daily as 2 separate doses.
  Open-label phase: Participants received ACR16 45 mg capsule once daily for the first 4 weeks (Weeks 26 to 30). After 4 weeks (Weeks 31 to 52), ACR16 45 mg capsule was taken twice daily as 2 separate doses (total dose: 90 mg).
- Total: Total of all reporting groups
Arm/Group | Placebo/ACR16 90 mg | ACR16 45 mg/90 mg | ACR16 90 mg/90 mg | Total
Number analyzed (Participants) | 144 | 148 | 145 | 437
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (9.6) | 51.0 (10.7) | 51.8 (11.1) | 50.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 82 | 64 | 222
  Male | 68 | 66 | 81 | 215
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 0 | 2 | 0 | 2
  Race: Other | 0 | 1 | 0 | 1
  Race: Caucasian | 144 | 145 | 145 | 434
Unified Huntington's Disease Rating Scale (UHDRS) Modified Motor Score (mMS) [Mean (Standard Deviation); unit: units on a scale] — The mMS is a subscale of the UHDRS total motor score and comprises 13 responses from the 10 items, 4-10 and 13-15, from the UHDRS motor assessment. The items for mMS included dysarthria, tongue protrusion, finger taps (right and left), pronate/supinate hands (right and left), luria - first-hand-palm sequencing, arms rigidity (right and left), body bradykinesia, gait, tandem walking, and retropulsion pull test. Each of these items were rated on a scale of 0 (normal) to 4 (marked impairment). Total score ranged from 0 to 52, with higher scores indicating more severe motor impairment.
  units on a scale | 19.43 (8.28) | 18.38 (6.76) | 18.57 (6.90) | 18.79 (7.34)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Motor Score (mMS) (Sum of Score of Items 4-10 and 13-15 of the Unified Huntington's Disease Rating Scale [UHDRS] Motor Assessments) at Week 26
Description: The mMS is a subscale of the UHDRS total motor score and comprises 13 responses from the 10 items, 4-10 and 13-15, from the UHDRS motor assessment. The items for mMS include dysarthria, tongue protrusion, finger taps (right and left), pronate/supinate hands (right and left), luria - first-hand-palm sequencing, arms rigidity (right and left), body bradykinesia, gait, tandem walking, and retropulsion pull test. Each of these items are rated on a scale of 0 (normal) to 4 (marked impairment). Total score ranges from 0 to 52, with higher scores indicating more severe motor impairment.
Time Frame: Baseline, Week 26
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug and had undergone at least 1 clinical assessment post randomization. Here, 'Overall number of participants analyzed signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo/ACR16 90 mg: Randomized phase: Participants received a placebo capsule matched to ACR16 once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 26), placebo capsule was taken twice daily as 2 separate doses.
  Open-label phase: Participants received ACR16 45 mg capsule once daily for the first 4 weeks (Weeks 26 to 30). After 4 weeks (Weeks 31 to 52), ACR16 45 mg capsule was taken twice daily as 2 separate doses (total dose: 90 mg).
- ACR16 45 mg/90 mg: Randomized phase: Participants received ACR16 45 milligrams (mg) capsule orally once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 26), one ACR16 45 mg capsule and one placebo capsule were taken as 2 separate doses.
  Open-label phase: Participants received ACR16 45 mg capsule once daily for the first 4 weeks (Weeks 26 to 30). After 4 weeks (Weeks 31 to 52), ACR16 45 mg capsule was taken twice daily as 2 separate doses (total dose: 90 mg).
Arm/Group | Placebo/ACR16 90 mg | ACR16 45 mg/90 mg | ACR16 90 mg/90 mg
Number analyzed (Participants) | 138 | 146 | 139
units on a scale | 0.27 (4.43) | -0.23 (4.12) | -0.94 (3.87)
Statistical Analysis 1: Comparison: Placebo/ACR16 90 mg vs ACR16 45 mg/90 mg; The analysis of covariance (ANCOVA) main effects model included a term for treatment and covariates for baseline mMS, gender, and use of antipsychotic medication; Test type: Superiority — This analysis compared ACR16 45 mg vs. placebo during the randomization phase; p = 0.456, ANCOVA; Mean Difference (Final Values) = -0.36, 97.5% CI 2-sided [-1.44 to 0.72]
Statistical Analysis 2: Comparison: Placebo/ACR16 90 mg vs ACR16 90 mg/90 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This analysis compared ACR16 90 mg vs. placebo during the randomization phase; p = 0.042, ANCOVA; Mean Difference (Final Values) = -0.99, 97.5% CI 2-sided [-2.08 to 0.10]

2. Secondary Outcome: The UHDRS Functional Assessment at Week 26
Description: The UHDRS Functional Assessment considers 25 items associated with functional problems. The participant scores 1 point for every item to which they respond positively (zero points for negative responses). Total score ranges from 0 (worst) to 25 (best). Higher scores indicate better functional ability.
Time Frame: Week 26
Population: FAS included all randomized participants who received at least 1 dose of study drug and had undergone at least 1 clinical assessment post randomization. Here, 'Overall number of participants analyzed signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo/ACR16 90 mg | ACR16 45 mg/90 mg | ACR16 90 mg/90 mg
Number analyzed (Participants) | 139 | 146 | 139
Units on a Scale | 16.81 (6.20) | 17.50 (5.73) | 17.48 (5.43)

3. Secondary Outcome: Number of Participants With Clinical Global Impression - Improvement (CGI-I) Score
Description: Global improvement is rated by the investigator on a 7-point scale as: 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = No change; 5 = Minimally worse; 6 = Much worse; and 7 = Very much worse.
Time Frame: Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/ACR16 90 mg | ACR16 45 mg/90 mg | ACR16 90 mg/90 mg
Number analyzed (Participants) | 139 | 146 | 140
Participants
  Very much improved | 1 | 1 | 1
  Much improved | 8 | 8 | 7
  Minimally improved | 30 | 32 | 33
  No change | 55 | 59 | 50
  Minimally worse | 38 | 37 | 46
  Much worse | 7 | 9 | 2
  Very much worse | 0 | 0 | 0
  Missing | 0 | 0 | 1

4. Secondary Outcome: Change From Baseline in Stroop Word Reading Test at Week 26
Description: The Stroop test measures the ability to concentrate and ward off distractions. The test consists of three items: (i) colour naming; (ii) word reading; (iii) interference. The word reading test requires participants to read colour words written in black and each response is scored as the number of correct answers made in 45 seconds. Higher scores indicate less severe disease, and an increase in score represents an improvement.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Placebo/ACR16 90 mg | ACR16 45 mg/90 mg | ACR16 90 mg/90 mg
Number analyzed (Participants) | 135 | 140 | 136
correct responses | -1.3 (11.9) | -1.1 (10.3) | -0.8 (11.7)

5. Secondary Outcome: Change From Baseline in Total UHDRS Behavioral Assessment Score at Week 26
Description: The total behavioral assessment score is the sum of the 11 products (depressed mood, apathy, low self-esteem/guilt, compulsive behavior, anxiety, irritable behavior, perseverative/obsessive thinking, disruptive/aggressive behavior, suicidal thoughts, delusions, and hallucinations) of frequency and severity symptom scores and excluded the 3 yes/no questions relating to confusion, dementia, and depression. Frequency is rated on a scale of 0 (never or almost never) to 4 (very frequently, most of the time). Severity is rated on a scale of 0 (no evidence) to 4 (severe). Total behavior score ranges from 0 (no impairment) to 88 (severe impairment), with higher scores indicating greater behavioral impairments.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/ACR16 90 mg | ACR16 45 mg/90 mg | ACR16 90 mg/90 mg
Number analyzed (Participants) | 139 | 146 | 139
units on a scale | 0.12 (13.51) | -0.41 (16.78) | -2.22 (10.84)

6. Secondary Outcome: Change From Baseline in Total Hospital Anxiety and Depression Scale (HADS) Score at Week 26
Description: HADS is a self-administered instrument reliable for detecting states of depression and anxiety. It includes 2 subscales: Hospital Anxiety and Depression Scale - anxiety (HADS-A) assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); Hospital Anxiety and Depression Scale - depression (HADS-D) assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale is comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score ranges from 0 to 21 for each subscale where higher scores indicate greater severity of anxiety and depression symptoms. The total HADS score was a composite score summed of all 14 items for a total range of 0 to 42. Lower change from baseline scores indicate improvement.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/ACR16 90 mg | ACR16 45 mg/90 mg | ACR16 90 mg/90 mg
Number analyzed (Participants) | 133 | 142 | 138
units on a scale | -0.10 (6.04) | -0.73 (6.78) | 0.13 (6.00)

7. Secondary Outcome: Randomized Phase: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any change from the participant's baseline (pre-treatment) condition, other than improvement, that did not necessarily have causal relationship with the study drug. TEAEs were defined as AEs that began after ACR16/placebo administration through week 26 or up to week 30 for participants not continuing in the open-label period. AEs included both serious adverse events (SAEs) and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline up to Week 30
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized Phase: Placebo: Participants received placebo matched to ACR16 in the randomized phase.
- Randomized Phase: ACR16 45 mg: Participants received ACR16 45 mg in the randomized phase.
- Randomized Phase: ACR16 90 mg: Participants received ACR16 90 mg in the randomized phase.
Arm/Group | Randomized Phase: Placebo | Randomized Phase: ACR16 45 mg | Randomized Phase: ACR16 90 mg
Number analyzed (Participants) | 144 | 148 | 145
Participants | 92 | 91 | 99

8. Secondary Outcome: Open-label Phase: Number of Participants With TEAEs
Description: An AE was defined as any change from the participant's baseline (pre-treatment) condition, other than improvement, that did not necessarily have causal relationship with the study drug. TEAEs were defined as adverse events that began after ACR16/placebo administration through Week 56. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Week 26 up to Week 56
Population: Open-label analysis set (OLAS) included the subset of participants who completed the randomized phase on study treatment and who consented to enter the open-label follow-up phase.
Measure: Count of Participants; unit: Participants
Groups:
- Open-label Phase: Placebo/ACR16 90 mg: Participants who received placebo during the randomized phase received ACR16 90 mg in the open-label phase.
- Open-label Phase: ACR16 45 mg/90 mg: Participants who received ACR16 45 mg during the randomized phase received ACR16 90 mg in the open-label phase.
- Open-label Phase: ACR16 90 mg/90 mg: Participants who received ACR16 90 mg during the randomized phase continued to receive ACR16 90 mg in the open-label phase.
Arm/Group | Open-label Phase: Placebo/ACR16 90 mg | Open-label Phase: ACR16 45 mg/90 mg | Open-label Phase: ACR16 90 mg/90 mg
Number analyzed (Participants) | 113 | 125 | 115
Participants | 90 | 101 | 95

ADVERSE EVENTS:
Time Frame: Baseline up to Week 56
Description: Safety set included all randomized participants who received at least 1 dose of study drug. The Open-label analysis set included participants who completed the randomized phase (RP) and entered the open-label phase (OLP). AEs were analyzed in the OLP for participants who received ACR16 in the RP and then received ACR16 90 mg in the OLP as one group combined per planned analysis. Participants who received placebo in the RP and received ACR16 90 mg in OLP were analyzed as a separate OL group.
Groups:
- Open Label Phase: Placebo: Participants who received placebo during the randomized phase and received ACR16 90 mg in the open label phase.
- Open Label Phase: ACR 16: Participants who received ACR16 45 mg or 90 mg in the randomized phase and received ACR16 90 mg in the open label phase.
Arm/Group | Randomized Phase: Placebo | Randomized Phase: ACR16 45 mg | Randomized Phase: ACR16 90 mg | Open Label Phase: Placebo | Open Label Phase: ACR 16
Serious Adverse Events (participants affected / at risk) | 11/144 | 10/148 | 9/145 | 6/113 | 15/240
Other Adverse Events (participants affected / at risk) | 54/144 | 49/148 | 56/145 | 38/113 | 88/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Phase: Placebo (N=144) | Randomized Phase: ACR16 45 mg (N=148) | Randomized Phase: ACR16 90 mg (N=145) | Open Label Phase: Placebo (N=113) | Open Label Phase: ACR 16 (N=240)
ANAL SPASM (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DISEASE PROGRESSION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FUME INHALATION DISORDER (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OVARIAN EPITHELIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AGGRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOKING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEURODERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HUNTINGTON'S CHOREA (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HELICOBACTER GASTRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GLASGOW COMA SCALE ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DUPUYTREN'S CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENTROPION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Phase: Placebo (N=144) | Randomized Phase: ACR16 45 mg (N=148) | Randomized Phase: ACR16 90 mg (N=145) | Open Label Phase: Placebo (N=113) | Open Label Phase: ACR 16 (N=240)
HUNTINGTON'S CHOREA (Congenital, familial and genetic disorders) | 9 (10) | 7 (7) | 10 (10) | 7 (7) | 29 (32)
DIARRHOEA (Gastrointestinal disorders) | 7 (8) | 10 (11) | 9 (10) | 3 (3) | 8 (9)
NAUSEA (Gastrointestinal disorders) | 9 (13) | 9 (11) | 5 (5) | 2 (2) | 5 (5)
FATIGUE (General disorders) | 9 (10) | 7 (8) | 4 (5) | 4 (4) | 6 (6)
NASOPHARYNGITIS (Infections and infestations) | 6 (6) | 9 (11) | 10 (10) | 5 (6) | 9 (10)
FALL (Injury, poisoning and procedural complications) | 12 (17) | 7 (10) | 15 (19) | 14 (14) | 24 (30)
DIZZINESS (Nervous system disorders) | 6 (6) | 10 (10) | 8 (18) | 4 (4) | 6 (7)
HEADACHE (Nervous system disorders) | 4 (5) | 4 (4) | 8 (8) | 4 (4) | 4 (4)
DEPRESSION (Psychiatric disorders) | 8 (8) | 6 (6) | 6 (6) | 4 (4) | 11 (11)
INSOMNIA (Psychiatric disorders) | 5 (5) | 5 (5) | 9 (11) | 3 (4) | 8 (8)
IRRITABILITY (General disorders) | 6 (6) | 3 (3) | 6 (6) | 6 (7) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 30 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.